CLINICAL TRIAL: NCT02316951
Title: Monitoring Postoperative Pain and Recovery Following Orthopedic Surgery
Status: Terminated | Type: Observational
Why Stopped: Logistical and enrollment issues
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400424
Record Dates: First submitted 2014-12-10; First posted 2014-12-15 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Pain, Postoperative
Keywords: Postoperative; Pain; Symptoms; Video recording; Orthopedic surgery
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single-arm study group: Study participants will be adult patients recovering from orthopedic surgery. The study group will wear a small motion detection device and a regular Webcam will be placed near the wall facing the bed in each patient's hospital room.
  Interventions: Device: single-arm study group

INTERVENTIONS:
Device: single-arm study group — Study participants will wear a small motion detection device and a regular Webcam will be placed near the wall facing the bed in each patient's hospital room. Study participants will be questioned about their sociodemographic, pain, and health history.

SUMMARY:
This pilot study will seek to use emotion recognition technology from video to link patient facial expressions, heart rate and respiratory rate changes, and movement patterns to patient pain scores.

DETAILED DESCRIPTION:
During hospitalization, beginning after orthopedic surgery, study participants will be asked to wear a small motion detector on their wrist. A computer vision system which analyzes both whole-body movement as well as facial expressions will be used at the bedside to compare common signs and symptoms of post op pain to patient pain scores.

Up to 30 study participants will be selected.

Study participants will be asked to complete a written pain diary during waking hours.This information will be compared to the pain scores found in the patient's medical record and/or the amount and frequency of pain medications they receive.

ELIGIBILITY:
Inclusion Criteria:

* Recovery following Orthopedic Surgery
* Non-vulnerable adult patient
* Residing on the 6th floor of the South Tower of UF Health Shands Hospital
* Under the care of the acute pain service

Exclusion Criteria:

* Inability to understand pain assessments
* Inability to wear a motion tracking device
* Amputation of limb
* Vulnerable subject status
* Anticipated discharge from hospital within 24 hours following enrollment
* < 21 years of age

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age >21) recovering from orthopedic surgery residing in an area hospital and under the care of the acute pain service.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2022-08-07 (Actual); Study Completion 2022-08-07 (Actual)

PRIMARY OUTCOMES:
pain assessment (Correlate pain scores with motion measurements obtained through measurement of movement activity and video.) | 1 day
  Correlate pain scores with motion measurements obtained through measurement of movement activity and video.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Tighe, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No